CLINICAL TRIAL: NCT04441645
Title: Effects of Acupressure Intervention on Cognitive Function and Quality of Life in Older Adults With Cognitive Impairment in Long-term Care Settings: A Cluster-Randomized Controlled Trial
Brief Title: Acupressure on Cognitive Function and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, I-Hui-Chen 陳逸卉, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 108MOST
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- the acupoint-on-head group (Experimental): pressing acupoints only on head
  Interventions: Other: Acupressure
- the acupoint-on-body group (Experimental): pressing acupoints only on body
  Interventions: Other: Acupressure
- the acupoint-on-head-and-body group (Experimental): pressing acupoints on head and body
  Interventions: Other: Acupressure
- the control group (No Intervention): routine care

INTERVENTIONS:
Other: Acupressure — acupressure once per day, five times per week, a total of 12 weeks
  Arms: the acupoint-on-body group; the acupoint-on-head group; the acupoint-on-head-and-body group

SUMMARY:
The study aims to (1)compare differences of global cognitive function, working memory, executive function, language function, and quality of life between institutionalized older adults with MCI and with mild AD. Doing so, we can have a better understanding of the cognitive performance and life quality at pre-dementia and dementia;(2)explore the effects of the interventions with different acupoints(acupoints on head, acupoints on body, and acupoints on head and body) on global cognitive function, working memory, executive function, language function, and quality of life among institutionalized older adults with MCI and with mild AD;(3) further investigate the long-term effects of the interventions on global cognitive function, working memory, executive function, language function, and quality of life among institutionalized older adults with MCI and with mild AD; doing this, we can explore the pathological mechanism of the changes in the cognitive function through neuropsychological assessments and the association between the changes in cognitive function and in quality of life. We will recruit 32 residential care homes, with 256 older adults with MCI and with mild AD for this single blind cluster randomized controlled trial with repeated measures study. The facilities will be randomly assigned to the acupoint-on-head group, acupoint-on-body group, acupoint-on-head-and-body group and control group, with a ratio of 1:1:1:1. Interventions are developed based on the theory of Chinese medicine. Except routine care, the intervention groups will receive the acupressure once per day, five times per week, a total of 12 weeks. Data will be collected at baseline, the 4th and 8th weeks during the intervention, the end of the intervention, and the1st, 4th, and 8th months after the intervention. The control group only will receive routine care and data collection is the same as the intervention groups. Data assessors will not involve in the interventions and not know the group allocation. The data analysis will use intent-to-treat analysis. The multiple regression analysis, mixed effect model for repeated measure analysis, subgroup analysis, and product-of-coefficient test will be performed to examine the effects of the interventions on cognitive function and quality of life, and the associations among the changes in the dependent variables.

DETAILED DESCRIPTION:
Although evidence has demonstrated that acupressure effectively improves older patients' symptoms (e.g., sleep disturbance, behavior and psychological symptoms of dementia, etc.), it is still lack of the study to investigate the effect of the acupressure on cognitive function and quality of life among older adults with cognitive impairment in long-term care settings and its long-term effects. In addition, according to statistical data for epidemiological investigation, the majority is people with mild cognitive impairment (MCI) and mild dementia (mild AD); hence, it is vital to prevent these two groups from having dementia or getting worse. The study aims to (1)compare differences of global cognitive function, working memory, executive function, language function, and quality of life between institutionalized older adults with MCI and with mild AD. Doing so, we can have a better understanding of the cognitive performance and life quality at pre-dementia and dementia;(2)explore the effects of the interventions with different acupoints(acupoints on head, acupoints on body, and acupoints on head and body) on global cognitive function, working memory, executive function, language function, and quality of life among institutionalized older adults with MCI and with mild AD;(3) further investigate the long-term effects of the interventions on global cognitive function, working memory, executive function, language function, and quality of life among institutionalized older adults with MCI and with mild AD; doing this, we can explore the pathological mechanism of the changes in the cognitive function through neuropsychological assessments and the association between the changes in cognitive function and in quality of life. This single blind cluster randomized controlled trial with repeated measures study will complete in 2 years. We will recruit 32 residential care homes in Taipei City, with 256 older adults with MCI and with mild AD. The facilities will be randomly assigned to the acupoint-on-head group, acupoint-on-body group, acupoint-on-head-and-body group and control group, with a ratio of 1:1:1:1. Interventions are developed based on the theory of Chinese medicine and the trained research assistants, also having traditional Chinese nursing training, will perform the interventions. Except routine care, the intervention groups will receive the acupressure once per day, five times per week, a total of 12 weeks. Data will be collected at baseline, the 4th and 8th weeks during the intervention, the end of the intervention, and the1st, 4th, and 8th months after the intervention. The control group only will receive routine care and data collection is the same as the intervention groups. Data assessors will not involve in the interventions and not know the group allocation. The data analysis will use intent-to-treat analysis. The multiple regression analysis, mixed effect model for repeated measure analysis, subgroup analysis, and product-of-coefficient test will be performed to examine the effects of the interventions on cognitive function and quality of life, and the associations among the changes in the dependent variables. This study will promote the professional nursing autonomy and improve life quality of the institutionalized older adults.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination (MMSE):20~28
* Clinical Dementia Rating (CDR): 0.5~1

Exclusion Criteria:

* CDR>1

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
The Cognitive Abilities Screening Instrument | up to 12 months
  a cognitive test screening for dementia in providing profiles of cognitive impairment by examining abilities on attention, concentration, orientation, short-term memory, long-term memory, language abilities, visual construction, list-generating fluency, abstraction, and judgment with score ranges of 0 to 100, respectively.

SECONDARY OUTCOMES:
The Digit Span Test | up to 12 months
  a key tool for working verbal memory.
The Wisconsin Card Sorting Test | up to 12 months
  a neuropsychological test of the ability to display flexibility in the face of changing schedules of reinforcement
Semantic Association of Verbal Fluency | up to 12 months
  the generation of words from a given category within a pre-set time of 60 seconds.
Quality of life-Alzheimer's disease scale | up to 12 months
  The QoL-AD is comprised of 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole). Response options include 1(poor), 2(fair), 3(good) and 4 (excellent), for a total score of 13-52, with higher scores indicating better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: I-Hui Chen, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan